CLINICAL TRIAL: NCT03691116
Title: Feasibility and Effectiveness of Digital Self-help Support for Lifestyle Behavior Changes Among Primary Care Outpatients With Mental Health Problems
Brief Title: Digital Self-help Support for Lifestyle Behavior Changes Among Primary Care Outpatients With Mental Health Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1013-31/4
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Mental Health; Risk Reduction Behavior; Primary Health Care
Keywords: Mental Health; Digital Intervention; Alcohol; Tobacco; Diet; Physical Activity; Primary Health Care
MeSH Terms: conditions — Psychological Well-Being; Risk Reduction Behavior; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Health Profile (Experimental): A digital health check-up, with questions, brief feedback and information about alcohol, tobacco, diet and exercise, as a complement to treatment as usual. (Psychological assessment and treatment)
  Interventions: Behavioral: Digital Health Profile; Behavioral: Treatment as usual
- Treatment as usual (Active Comparator): Psychological assessment and treatment as usual.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Digital Health Profile — Screening, health check-up and automatic feedback in the areas tobacco, alcohol, exercise and diet, used on a National digital platform (Stöd och Behandlingsplattformen, SoB)
  Arms: Digital Health Profile
Behavioral: Treatment as usual — Ordinary psychological assessment and counseling.

SUMMARY:
All patients, who have booked a first appointment with a psychologist or counselor at two primary care clinics, are asked to fill out a lifestyle screening questionnaire within the Electronic Medical Record (EMR) system. Up to 150 patients will be screened. The patients who have filled out the first screening and given informed consent are randomized to either Group A: A digital health check-up, with more questions and brief feedback; or Group B: Treatment as usual.

The digital health check-up is based on "Hälsoprofilen", a material that successfully has been used with thousands of patients in Western Sweden. This material generates brief feedback to the patients about the status of their lifestyle behavior and indicates the need for change when necessary for better health. After 10 weeks, the patients fill in the first short screening again. Outcome analyses will compare the two groups.

DETAILED DESCRIPTION:
The study will be carried out at two primary care clinics in Stockholm. All patients, who have booked a first appointment with a psychologist or counselor at two primary care clinics, are asked to fill out a lifestyle screening questionnaire within the Electronic Medical Record (EMR) system. Up to 150 patients will be screened. The patients who have filled out the first screening and given informed consent are randomized to either Group A: A digital health check-up, with more questions and brief feedback; or Group B: Treatment as usual.

The digital health check-up is based on "Hälsoprofilen", a material that successfully has been used with thousands of patients in Western Sweden. This material generates brief feedback to the patients about the status of their lifestyle behavior and indicates the need for change when necessary for better health. After 10 weeks, the patients fill in the first short screening again. Outcome analyses will compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients that seeks psychological treatment during the time period when the study is ongoing.

Exclusion Criteria:

* Children under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 10 weeks
  Self administered depression scores
Generalized Anxiety Disorder (GAD-7) | 10 weeks
  Self administered anxiety scores

SECONDARY OUTCOMES:
Lifestyle habits | 10 weeks
  Self administered lifestyle scores,

OTHER OUTCOMES:
Feasibility assessment | 10 weeks
  Mapping participant lifestyle habits and evaluating whether the model works in ordinary primary care setting.
  Assessed via patient and staff interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Liljeholmens Primary Healthcare Center, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolaas K, Axelsson E, Hedman-Lagerlof E, Berman AH. Healthy lifestyle promotion via digital self-help for mental health patients in primary care: a pilot study including an embedded randomized recruitment trial. Prim Health Care Res Dev. 2023 Sep 20;24:e56. doi: 10.1017/S146342362300049X. PMID 37728142